CLINICAL TRIAL: NCT05496101
Title: Intraoperative Assessment of Tumour Excision Margins Using the LightPath Imaging System for Cerenkov Luminescence Imaging (CLI) Combined With Flexible Autoradiography (FAR) in Women Undergoing Breast-conserving Surgery (BCS)
Brief Title: CLI and FAR for Intraoperative Margin Assessment
Acronym: CLI-FAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 314460
Record Dates: First submitted 2022-04-29; First posted 2022-08-11 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Intervention Model Description: Intraoperative CLI + FAR LightPath imaging with comparator-Standard-of-care histopathology (gold standard)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast Cancer undergoing BCS (Other): Intraoperative CLI + FAR LightPath imaging compared with Standard-of-care histopathology (gold standard)
  Interventions: Procedure: Intraoperative CLI + FAR LightPath imaging

INTERVENTIONS:
Procedure: Intraoperative CLI + FAR LightPath imaging — Imaging System: The LightPath Imaging System is an in vitro diagnostic device which has CE mark in Europe, in line with In Vitro Diagnostic Medical Devices 98/79/EC (post marketing study).
  Radiopharmaceutical:
  18F-FDG is a routinely used Positron Emission Tomography (PET) / Computed Tomography (CT) radiopharmaceutical

SUMMARY:
This study is a prospective, single arm interventional study to evaluate the diagnostic accuracy of intraoperative Cerenkov luminescence imaging (CLI) plus flexible autoradiography (FAR) using the LightPath® Imaging System for intraoperative tumour margin assessment compared to post-operative standard-of-care histopathology in women undergoing breast-conserving surgery for breast cancer.

DETAILED DESCRIPTION:
The intraoperative LightPath images will be used to inform the operating surgeon about potentially detectable cancer at the margins of the excised specimen in an attempt to achieve better guided cancer surgery and complete tumour excision with clear resection margins. If a positive excision margin is detected on intraoperative LightPath® images, the operating surgeon will take a cavity shaving of the corresponding margin, provided more tissue can be taken. Subsequent LightPath® imaging of the cavity shaving will inform the operating surgeon on the margin status of the shaving. If a positive excision margin is detected on intraoperative LightPath® images, the operating surgeon will take a further cavity shave of the corresponding margin, provided more tissue can be taken.

The resection margin status of the WLE specimen and cavity shavings (if any), as assessed by LightPath CLI + FAR imaging will be compared with final histopathology results.

A positive margin on histology will be defined as

* Invasive carcinoma: positive: <1mm; negative ≥1mm
* Ductal carcinoma in situ (DCIS) (if present): positive: <2mm; negative ≥2mm.

ELIGIBILITY:
Inclusion Criteria:

* • Female subjects ≥18 years of age with a diagnosis of invasive breast cancer scheduled to undergo BCS

  * Subjects who are able to give voluntary, written informed consent to participate in this study
  * Subjects who are able to understand this study and are willing to complete all the study assessments
  * Female subjects of childbearing age must have a negative pregnancy test (by Beta human chorionic gonadotrophin (β-HCG) qualitative analysis) or must have had a history of a surgical sterilisation or must give history of no menses in the past twelve months.

Exclusion Criteria:

* Subjects who have had surgery to the ipsilateral breast in the past 12 months
* Subjects who have had radiotherapy to the ipsilateral breast
* Subjects who have a known hypersensitivity to 18F-FDG
* Subjects who are pregnant or lactating
* Subjects who have an existing medical condition that would compromise their participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological representation
Enrollment: 60 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Margin status of WLE specimens | complete surgical procedure
  The resection margin status of the WLE specimen and cavity shavings (if any), as assessed by LightPath CLI + FAR imaging will be compared with final histopathology results. A positive margin on histology will be defined as
  * Invasive carcinoma: positive: <1mm; negative ≥1mm
  * Ductal carcinoma in situ (DCIS) (if present): positive: <2mm; negative ≥2mm. The resection margin status of the WLE specimen and cavity shavings (if any), as assessed by LightPath CLI + FAR imaging will be compared with final histopathology results. A positive margin on histology will be defined as
  * Invasive carcinoma: positive: <1mm; negative ≥1mm
  * Ductal carcinoma in situ (DCIS) (if present): positive: <2mm; negative ≥2mm.

SECONDARY OUTCOMES:
• Agreement between margin status of cavity shavings as determined by intraoperative CLI + FAR LightPath imaging and post-operative histopathology. | complete surgical procedure
  • Re-operation rate within the study cohort compared to general breast cancer population undergoing a WLE.

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No